CLINICAL TRIAL: NCT00021346
Title: Phase I Evaluation Of Carboplatin And Gemcitabine
Brief Title: Carboplatin and Gemcitabine in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068771; P30CA006927 (NIH); FCCC-97028; NCI-G01-1984
Record Dates: First submitted 2001-07-11; First posted 2004-04-22 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Carboplatin; Gemcitabine

INTERVENTIONS:
Drug: carboplatin
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining carboplatin and gemcitabine in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of gemcitabine and carboplatin in patients with advanced solid tumors. II. Determine the dose-limiting toxic effects of this regimen in these patients. III. Evaluate the pharmacokinetics and pharmacodynamics of this regimen in these patients. IV. Determine the observed responses in these patients receiving this regimen.

OUTLINE: This is a dose-escalation study of gemcitabine. Patients are stratified according to prior therapy (no prior chemotherapy and/or prior radiotherapy to less than 20% of bone marrow vs prior chemotherapy and/or prior radiotherapy to at least 20% of bone marrow). Patients receive carboplatin IV over 30 minutes on day 1 and gemcitabine IV over 30 minutes on days 1 and 8. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity. Cohorts of 1-3 patients receive escalating doses of gemcitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 patients experience dose-limiting toxicity. Patients are followed for survival.

PROJECTED ACCRUAL: A maximum of 18 patients (9 per stratum) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed advanced solid tumor for which no standard therapy exists No untreated brain metastases with evidence of neurologic deterioration or CNS progression

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-1 Life expectancy: More than 3 months Hematopoietic: Absolute neutrophil count at least 2,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL SGOT no greater than 5 times upper limit of normal Renal: Creatinine no greater than 1.5 mg/dL Other: No serious concurrent infection No other serious concurrent medical illness that would preclude study Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for at least 3 months after study

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No more than 2 prior systemic chemotherapy regimens for advanced disease Prior adjuvant or induction therapy for initial disease allowed At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas, mitomycin, or melphalan) No prior combination carboplatin and gemcitabine Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy to more than 30% of bone marrow At least 4 weeks since prior radiotherapy Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 1997-11; Primary Completion 2001-07 (Actual); Study Completion 2002-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corey J. Langer, MD, Study Chair — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States